CLINICAL TRIAL: NCT02318121
Title: Concurrent Versus Sequential Administration of Amniotomy and Oxytocin for Augmentation of Labour: a Randomized Controlled Trial
Brief Title: Amniotomy and Oxytocin for Augmentation of Labour
Acronym: AOAL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Omar Mamdouh Shaaban, Dr., Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Augmentation of labour
Record Dates: First submitted 2014-10-05; First posted 2014-12-17 (Estimated); Last update posted 2017-11-21 (Actual); Status verified 2017-11

CONDITIONS: Prolonged Labor
Keywords: Labor, prolonged labor, augmentation of labor
MeSH Terms: interventions — Amniotomy; Oxytocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Amniotomy first (Active Comparator): Will be done with sterile gloves after insurance that is the baby's head fits in the pelvis ( 3\5 or less of fetal head felt by first pelvic grip ) and by vaginal examination the head at station zero . The membranes are then punctured using an a hook during uterine contractions.
  Interventions: Procedure: Amniotomy first
- Oxytocin first (Active Comparator): The starting dose will be the low dose rate equal or less than 4 m unit\minute (4 drops\minute doubled every 15 minutes up to 40 drops \minute) as intravenous drip on dextrose ,Ringer's lactate or saline solution.
  Interventions: Procedure: Oxytocin first; Drug: Oxytocin
- Amniotomy and oxytocin (Active Comparator): Amniotomy will be done (as explained above) and oxytocin (the same regimen mentioned above) at the same time.
  Interventions: Procedure: Amniotomy and oxytocin; Drug: Oxytocin

INTERVENTIONS:
Procedure: Amniotomy first — rupture of membranes to augment labor
  Arms: Amniotomy first
Procedure: Oxytocin first — Administration of oxytocin to augment labor
  Arms: Oxytocin first
Procedure: Amniotomy and oxytocin — Rupture of membranes and administration of oxytocin to augment labor
  Arms: Amniotomy and oxytocin
Drug: Oxytocin
  Arms: Amniotomy and oxytocin; Oxytocin first

SUMMARY:
Prolonged labour is a cause of maternal mortality and morbidity and perinatal mortality and morbidity. Prolonged labour is most often defined as onset of regular , rhythmical painful contractions accompanied by cervical dilatation where labour is longer than 24 hours.prolonged active phase should not last longer than 12 hours without full assessment in a facility able to offer management and treatment of complications.Causes of prolonged labour usually due to poor or uncoordinated uterine action , fetal head malposition , and or abnormal pelvis either due to bone or soft tissue obstruction.

Arrested or prolonged labor is a frequent indication of cesarean delivery.Prolonged labor is also associated with increased pain and negative birth experience. Women with a prolonged first stage of labor have experienced a higher rate of postpartum hemorrhage, chorioamnionitis and neonatal admission to the intensive care unit.

Caesarean section rates are over 20% in many developed countries and have increased nearly four-fold relative to the 5% rate observed in the early 1970s. The main diagnosis contributing to this increase is dystocia or prolonged labor.Data obtained from local hospital records showed that Caesarean section rate in Assiut University Women's Health Hospital is 47.96% at 2013.

Dystocia is a term used for delay of labor progress and usually refers to abnormally slow cervical dilatation.It has been proposed that the partogram should include, as a diagnostic criterion, a 1 cm/hour line originating at admission. The World Health Organization has proposed a modified partogram that recommends that active phase be diagnosed only at 4 cm or more.

Oxytocin augmentation of uterine contractions with or without amniotomy is widely used in the modern obstetric practice to treat a slow labour, although the timing of oxytocin initiation and amniotomy may vary widely.This intervention is based on the hypothesis that the most frequent cause of dystocia is inadequate uterine contraction.

The mechanism by which amniotomy speeds up labour remains unclear it is thought that when the membranes are ruptured ,the production and release of prostaglandins and oxytocin increases resulting in stronger contractions and quicker cervical dilatation. I has been found that early intervention (augmentation versus routine care ) with amniotomy and oxytocin to be associated with a modest reduction in the risk of caesarean section. Moreover, amniotomy found to be associated with an increased risk of cesarean delivery compared with women without amniotomy for shortening of spontaneous labour.

The 3 methods ( Amniotomy, Oxytocin or both) used for augmentation of labor in different settings without a real conclusion which is better.

ELIGIBILITY:
Inclusion Criteria:

* Women in spontaneous labor
* Women with intact membranes at the time of randomization
* Single fetus
* Vertex presentation
* Cervical dilatation 3 cm or more
* Gestational age 37 weeks or more proved by reliable dates or by early ultrasound scan in the first trimester
* Slow progress in the active phase of labor ( cervical dilatation less than 1 cm \hour)

Exclusion Criteria:

* Women with a previous uterine scar
* Severe preeclamptic toxemia
* Suspected fetal macrosomia (greater than 4000 g)
* Women with any congenital malformations
* Women with Intra uterine fetal death
* Diabetes mellitus with pregnancy
* Antepartum hemorrhage
* Women with other indications of caesarean section

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2014-04-01; Primary Completion 2014-09-01 (Actual); Study Completion 2015-12-01 (Actual)

PRIMARY OUTCOMES:
Rate of cervical dilatation | every hour up to full cervical dilatation
  The rate of cervical dilation cm/ hour

SECONDARY OUTCOMES:
Augmentation delivery time | Time ( in minutes) between the start of augmentation of labor up to the delivery of the head
  the duration between Augmentation of labor and the end of the second stage if labor
Apgar score at 10 minutes | from 0-10 minutes
  Assessment of Apgar score of the baby at 10 minutes after delivery